CLINICAL TRIAL: NCT05578482
Title: The Pathogenic Role Of Staphylococcus Aureus And The Skin Microbiome During Flare And Resolution Of Atopic Dermatitis
Brief Title: Staphylococcus Aureus and The Skin Microbiome During Flare And Resolution Of Atopic Dermatitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jacob Pontoppidan Thyssen (Other)
Collaborators: The Novo Nordic Foundation (Other)
Responsible Party: Sponsor-Investigator, Jacob Pontoppidan Thyssen, Professor, Jacob Pontoppidan Thyssen, Bispebjerg Hospital
Organization: Bispebjerg Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AR-AB-AD; 2021-006883-25 (EudraCT Number)
Record Dates: First submitted 2022-09-30; First posted 2022-10-13 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Atopic Dermatitis; Atopic Dermatitis Eczema; Atopic Dermatitis Flare
Keywords: Atopic dermatitis; Atopic dermatitis flare; Skin microbiome; Skin barrier markers; RCT; Antibiotics; Topical corticosteroids; Staphylococcus aureus
MeSH Terms: conditions — Dermatitis, Atopic; Staphylococcal Infections | interventions — Dicloxacillin; Mometasone Furoate

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial, Double Blinded
Who Masked: Participant, Investigator
Masking Description: The investigators as well as the participating patients are blinded during the RCT of Dicloxacillin/Placebo & Elocon
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dicillin & Elocon (Active Comparator): 20 of the participating patients are randomized to the active arm where systemic dicloxacillin and elocon creme (mometasone furoate 0.1%) is received.
  Interventions: Drug: Dicloxacillin Oral Capsule; Drug: Elocon 0.1 % Topical Cream
- Placebo & Elocon (Placebo Comparator): 20 of the participating patients are randomized to the placebo arm where placebo and elocon creme (mometasone furoate 0.1%) is received.
  Interventions: Drug: Elocon 0.1 % Topical Cream

INTERVENTIONS:
Drug: Dicloxacillin Oral Capsule — Randomized to either systemic dicloxacillin & elocon or placebo & elocon
  Other Names: Elocon (Mometasone furoate 0.1%)
  Arms: Dicillin & Elocon
Drug: Elocon 0.1 % Topical Cream — Both groups are treated with elocon for five days.
  Other Names: Mometasone furoate 0.1%

SUMMARY:
The goal of this clinical trial is to compare and evaluate in patients with atopic dermatitis. The main questions it aims to answer are:

* Does the addition of systemic dicloxacillin to TCS treatment result in a more rapid and deeper treatment response?
* Does the addition of systemic dicloxacillin to TCS treatment affect the skin microbiome, the skin barrier and immune response during improvement of AD?
* Does topical application of S. aureus or SEB increase the severity and rapidity of a flare?

Participants will meet for two different phases:

* Phase one will be at randomized controlled trial where patients are randomized to either systemic dicloxacillin + mometasone furoate or placebo + mometasone furoate.
* Phase II: Patients will meet for five visits to receive different solutions on the skin including autologous s. aureus and staphylococcal enterotoxin B.

DETAILED DESCRIPTION:
The investigators hypothesize:

Use of oral systemic antibiotic treatment with dicloxacillin (1000 mg x 3 times a day) will decrease the time to AD improvement as well as the amount of S. aureus and its toxins and alter the skin microbiome.

Specifically, the investigators aim to investigate the following research questions:

* RQ1: Does the addition of systemic dicloxacillin to TCS treatment result in a more rapid and deeper treatment response?
* RQ2: Does the addition of systemic dicloxacillin to TCS treatment affect the skin microbiome, the skin barrier and immune response during improvement of AD?
* RQ3: Does topical application of S. aureus or SEB increase the severity and rapidity of a flare?
* RQ4: Does topical application of S. aureus and SEB alter the skin microbiome, the skin barrier and immune response during a flare of AD?
* RQ5: Can changes in protein expression or metabolic pathways explain the modulated mechanisms in the host-microbial cross talk of AD?

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or above
* European ancestry
* AD diagnosis according to Hanifin & Rajka criteria
* AD for at least 3 years
* AD that is moderate-to-severe defined as an EASI score of ≥ 7
* AD in the sampled location that has an TLSS score of ≥ 5

EXCLUSION CRITERIA:

* Current or present systemic immunosuppressant and/or biological treatment for the past 4 weeks
* Evidence of other concomitant inflammatory skin conditions (e.g., psoriasis or contact dermatitis)
* Evidence of active skin infection that warrants treatment at screening or baseline visit
* Systemic or topical antibiotics in the preceding past 4 weeks
* Use of disinfectants, bleach and potassium permanganate baths at least 2 weeks before sampling
* UV therapy within the last 3 weeks, or pronounced exposure to sunlight in the preceding 2 weeks
* History of any condition (e.g. bleeding diathesis) that may predispose the patient to complications associated with the planned skin biopsy procedures
* Other clinically significant medical disease that is uncontrolled despite treatment that is likely, in the opinion of the investigator, to impact the patient's ability to participate in the study or to impact the study pharmacodynamic, or safety assessments
* Decreased kidney function (GFR under 60 ml/min)
* Tendency to formation of keloid scars
* Penicillin or mometasone futurate allergy or intolerance
* Pregnancy
* Breast feeding
* Body weight ≤ 40 kg
* AD only located in the face or intimate regions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-10-24 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Change in The Total Lesion Symptom Scale (TLSS) score improvement | Through study completion, an average of 1 year
  The primary endpoint is to describe if addition of systemic dicloxacillin treatment (1000 mg x 3 times a day) to topical treatment with mometasone furoate 0.1% cream once daily increases the rapidity and depth of the treatment response measured as changes in The Total Lesion Symptom Scale (TLSS) score improvement. The score is a numerical scale from 0-15.

SECONDARY OUTCOMES:
Changes in the skin microbiome measured as community composition (beta-diversity) visualised as PCOA plots | 1 year
  Describe changes in the skin microbiome measured as community composition during i) treatment with systemic dicloxacillin treatment (1000 mg x 3 times a day) and mometasone furoate 0.1% cream once daily ii) treatment with mometasone furoate 0.1% cream once daily iii) cutaneous application of respectively SEB and S. aureus from the patient's self, compared to vehicle
Changes in the skin microbiome measured as alfa-diversity (Shannon diversity) | 1 year
  Describe changes in the skin microbiome measured as immune response during i) treatment with systemic dicloxacillin treatment (1000 mg x 3 times a day) and mometasone furoate 0.1% cream once daily ii) treatment with mometasone furoate 0.1% cream once daily iii) cutaneous application of respectively SEB and S. aureus from the patient's self, compared to vehicle
Changes in the skin microbiome measured as relative abundance (%) of baterial genera | 1 year
  During i) treatment with systemic dicloxacillin treatment (1000 mg x 3 times a day) and mometasone furoate 0.1% cream once daily ii) treatment with mometasone furoate 0.1% cream once daily iii) cutaneous application of respectively SEB and S. aureus from the patient's self, compared to vehicle
Changes in the amount of cytokines | 1 year
  Describe changes in the epidermal barrier disruption through changes in cytokines (to Il-1a, IL-4, IL-13, IL-1RA, CXCL-9, IL-22, IL-31, IL-8, IL-18, CCL-17, CCL-18, CCL-20, CCL-22, CXCL-10, VEGF-A) during i) treatment with systemic dicloxacillin treatment (1000 mg x 3 times a day) and mometasone furoate 0.1% cream once daily ii) treatment with mometasone furoate 0.1% cream once daily iii) cutaneous application of respectively SEB and S. aureus from the patient's self, compared to vehicle
Changes in itch with peak pruritus 24 hours | Through study completion, an average of 1 year
  Changes in itch on a scale from 0-10 during i) treatment with systemic dicloxacillin treatment (1000 mg x 3 times a day) and mometasone furoate 0.1% cream once daily ii) treatment with mometasone furoate 0.1% cream once daily iii) cutaneous application of respectively SEB and S. aureus from the patient's self, compared to vehicle.
The effects of treatment on markers of bone resorption and formation with C-terminal telopeptide of type I collagen (CTX) | 1 year
  The investigators aim to investigate the effects of treatment on markers of bone resorption and formation including C-terminal telopeptide of type I collagen (CTX) because TCS such as mometasone furoate may increase bone resorption as seen in a large epidemiologic study.
The effects of treatment on markers of bone resorption and formation with N-terminal propeptide of type 1 procollagen (P1NP) | 1 year
  The investigators aim to investigate the effects of treatment on markers of bone resorption and formation including N-terminal propeptide of type 1 procollagen (P1NP) because TCS such as mometasone furoate may increase bone resorption as seen in a large epidemiologic study.
The effects of treatment on markers of bone resorption and formation with parathyroid hormone (PTH) | 1 year
  The investigators aim to investigate the effects of treatment on markers of bone resorption and formation including parathyroid hormone (PTH), because TCS such as mometasone furoate may increase bone resorption as seen in a large epidemiologic study.
Changes in sleep-Numeric rating scale | Through study completion, an average of 1 year
  Changes in sleep on a numerical rating scale from 0-10 during: i) treatment with systemic dicloxacillin treatment (1000 mg x 3 times a day) and mometasone furoate 0.1% cream once daily ii) treatment with mometasone furoate 0.1% cream once daily iii) cutaneous application of respectively SEB and S. aureus from the patient's self, compared to vehicle.
Changes in pain-Numeric rating scale | Through study completion, an average of 1 year
  Changes in pain on a numerical rating scale from 0-10 during: i) treatment with systemic dicloxacillin treatment (1000 mg x 3 times a day) and mometasone furoate 0.1% cream once daily ii) treatment with mometasone furoate 0.1% cream once daily iii) cutaneous application of respectively SEB and S. aureus from the patient's self, compared to vehicle.
The Eczema Area and Severity Index (EASI) | Through study completion, an average of 1 year
  Changes in EASI score during: i) treatment with systemic dicloxacillin treatment (1000 mg x 3 times a day) and mometasone furoate 0.1% cream once daily ii) treatment with mometasone furoate 0.1% cream once daily iii) cutaneous application of respectively SEB and S. aureus from the patient's self, compared to vehicle.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Thyssen, Professor, MD, DMSc, Principal Investigator — Professor, Department of Dermatology, Bispebjerg Hospital
Locations (1):
- Department of Dermatology, Copenhagen NV, Denmark

IPD SHARING:
Plan to Share IPD: No
Due to Danish data protection law sharing IPD is not planned. Data outcomes should be anonymized without any recognizable information.

REFERENCES:
- [Derived] Ronnstad ATM, Bay L, Ruge IF, Halling AS, Fritz BG, Jakasa I, Luiten R, Kezic S, Thomsen SF, Bjarnsholt T, Thyssen JP. Defining the temporal relationship between the skin microbiome, immune response and skin barrier function during flare and resolution of atopic dermatitis: protocol of a Danish intervention study. BMJ Open. 2023 Feb 17;13(2):e068395. doi: 10.1136/bmjopen-2022-068395. PMID 36806068